CLINICAL TRIAL: NCT03094702
Title: Influence of SPRINT Trial Type Blood Pressure Measurements on Hypertension Diagnosis in Patients After Kidney Transplantation
Brief Title: SPRINT Trial Type Blood Pressure Measurements in Patients After Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Matthias Girndt, Director of the Department of Internal Medicine II, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: UKH-KIMII-001-17
Record Dates: First submitted 2017-03-09; First posted 2017-03-29 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Arterial Hypertension; Kidney Transplant; Complications
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SPRINT study used a blood pressure measurement procedure that differs from earlier studies in arterial hypertension. SPRINT type readings are lower than regular office measurements. The extent of the disagreement between SPRINT and office measurements may differ in distinct patient groups. This difference is not yet known for patients after renal transplantation. However, it is important to know the difference in order to apply SPRINT findings to transplant recipients.

DETAILED DESCRIPTION:
Most clinical trials on the treatment of arterial hypertension use office blood pressure measurements (Franklin et al. 2001; Hansson et al. 1998) both as inclusion criteria and study end-points. In these trials, blood pressure is taken by manual or automated devices in outpatients coming to a study center, as recommended by the European Society of Cardiology/European Society of Hypertension (ESC/ESH) Guidelines for the management of arterial hypertension (Mancia et al. 2013). The target blood pressure as recommended by European (Mancia et al. 2013) or US (James et al. 2014) guidelines largely depends on the results of the Hypertension Optimal Treatment (HOT) study (Hansson et al. 1998). This large trial with >18.000 participants measured blood pressure with an oscillometric device three times in a row in seated patients after 5min of rest. This and similar trials form the backbone of our knowledge about what is considered normal blood pressure and what blood pressure levels should be aimed at when using antihypertensive treatment (Zanchetti et al. 2009).

Studies using 24h-blood pressure measurement devices indicated that the normal values are lower (average 10/5mmHg) with this technique than with regular office measurements (Head et al. 2010). It is well known that there is a so called "white coat" hypertension, i.e. higher blood pressure values are taken in the doctor's office than at home (Mancia et al. 1987). The amount of this white-coat effect is largely different between individuals. Although white-coat hypertension itself has some prognostic impact on the patient (Verdecchia et al. 2005) it is much less relevant than overt hypertension. It seems reasonable to keep the White coat effect in mind to avoid over-therapy in patients in whom this effect is particularly strong.

While the framework for clinical decision making is mostly based on studies using office blood pressure readings, the SPRINT study (Wright et al. 2015) recently used another way of measuring blood pressure. The SPRINT study included more than 9.300 cardiovascular high-risk individuals without diabetes mellitus. It was a randomized prospective trial with intervention aiming at a low (<120 mmHg) vs. standard (<140 mmHg) systolic blood pressure. The trial was stopped early because of the large benefit of the intervention on the combined cardiovascular end-point. Since publication of this study, there is a vivid scientific discussion whether the low blood pressure goal should be aimed at in different patient populations.

The SPRINT study used a unique way of determining blood pressure. Patients were left alone in a quiet room with a programmed blood-pressure reading device that took readings at intervals after 5 minutes of relaxing. Recent studies showed that the blood pressure readings taken with the SPRINT technique are relevantly lower than the readings with regular office blood pressure measurements (Wohlfahrt et al. 2016).

Patients after renal transplantation very frequently have arterial hypertension (Kasiske et al. 2004; Paoletti et al. 2009). This is in part induced by the kidney disease or effects of the transplant and the immunosuppressive therapy; thus it might be considered a form of secondary hypertension. The KDIGO guideline (KDIGO clinical practice guideline for the care of kidney transplant recipients 2009) recommends to maintain blood pressure <130/80 mmHg in these patients. This recommendation is based on analogy to data from the general population and has not been formally proven in transplant patients. In order to determine if the SPRINT results can be extrapolated to transplant recipients as well, it is important to show the effect size of the different blood pressure measurement techniques (SPRINT vs. regular office BP) in this particular patient group.

The study intends to quantify the difference in blood pressure when read by regular ("real life") measurement or by the SPRINT procedure (primary goal).

In addition the study will describe factors that influence this difference (e.g. renal function, proteinuria, age, time since transplantation...) (secondary goals).

ELIGIBILITY:
Inclusion Criteria:

* Patients (m/f) with a functional renal transplant who are not dependent on dialysis treatment
* Age 18 - 99 years
* Riva-Rocchi blood pressure measurement at least at one arm possible
* Informed consent

Exclusion Criteria:

* No consent with study participation
* Psychiatric disorders preventing from valid informed consent
* Pregnancy or lactation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients (m/f) with a functional renal transplant who are not dependent on dialysis treatment
  * Age 18 - 99 years
  * Riva-Rocchi blood pressure measurement at least at one arm possible
  * Informed consent
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Difference between Office Blood Pressure and SPRINT type BP | Single Measurement at inclusion (day 1)
  Manual Office blood pressure [mmHg] minus Automated Office blood pressure [mmHg]

SECONDARY OUTCOMES:
Renal Function | Single Measurement at inclusion (day 1)
  Estimated Glomerular Filtration Rate (eGFR) [ml/min]
Proteinuria | Single Measurement at inclusion (day 1)
  Albumin-Creatinine-Ratio [g/g] or Protein concentration in 24h collected Urine [mmol/l]
Immunosuppressant use | Data acquisition at inclusion (day 1)
  Dose of Immunosuppression given as ddd [daily defined doses]

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Girndt, Prof. Dr., Study Chair — Department of Internal Medicine II, Martin-Luther-Universität Halle-Wittenberg
Locations (1):
- Internal Medicine II, Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Franklin SS, Larson MG, Khan SA, Wong ND, Leip EP, Kannel WB, Levy D. Does the relation of blood pressure to coronary heart disease risk change with aging? The Framingham Heart Study. Circulation. 2001 Mar 6;103(9):1245-9. doi: 10.1161/01.cir.103.9.1245. PMID 11238268
- [Background] Hansson L, Zanchetti A, Carruthers SG, Dahlof B, Elmfeldt D, Julius S, Menard J, Rahn KH, Wedel H, Westerling S. Effects of intensive blood-pressure lowering and low-dose aspirin in patients with hypertension: principal results of the Hypertension Optimal Treatment (HOT) randomised trial. HOT Study Group. Lancet. 1998 Jun 13;351(9118):1755-62. doi: 10.1016/s0140-6736(98)04311-6. PMID 9635947
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Zanchetti A, Grassi G, Mancia G. When should antihypertensive drug treatment be initiated and to what levels should systolic blood pressure be lowered? A critical reappraisal. J Hypertens. 2009 May;27(5):923-34. doi: 10.1097/HJH.0b013e32832aa6b5. PMID 19381107
- [Background] Head GA, Mihailidou AS, Duggan KA, Beilin LJ, Berry N, Brown MA, Bune AJ, Cowley D, Chalmers JP, Howe PR, Hodgson J, Ludbrook J, Mangoni AA, McGrath BP, Nelson MR, Sharman JE, Stowasser M; Ambulatory Blood Pressure Working Group of the High Blood Pressure Research Council of Australia. Definition of ambulatory blood pressure targets for diagnosis and treatment of hypertension in relation to clinic blood pressure: prospective cohort study. BMJ. 2010 Apr 14;340:c1104. doi: 10.1136/bmj.c1104. PMID 20392760
- [Background] Mancia G, Parati G, Pomidossi G, Grassi G, Casadei R, Zanchetti A. Alerting reaction and rise in blood pressure during measurement by physician and nurse. Hypertension. 1987 Feb;9(2):209-15. doi: 10.1161/01.hyp.9.2.209. PMID 3818018
- [Background] Verdecchia P, Reboldi GP, Angeli F, Schillaci G, Schwartz JE, Pickering TG, Imai Y, Ohkubo T, Kario K. Short- and long-term incidence of stroke in white-coat hypertension. Hypertension. 2005 Feb;45(2):203-8. doi: 10.1161/01.HYP.0000151623.49780.89. Epub 2004 Dec 13. PMID 15596572
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Wohlfahrt P, Cifkova R, Movsisyan N, Kunzova S, Lesovsky J, Homolka M, Soska V, Bauerova H, Lopez-Jimenez F, Sochor O. Threshold for diagnosing hypertension by automated office blood pressure using random sample population data. J Hypertens. 2016 Nov;34(11):2180-6. doi: 10.1097/HJH.0000000000001076. PMID 27512968
- [Background] Kasiske BL, Anjum S, Shah R, Skogen J, Kandaswamy C, Danielson B, O'Shaughnessy EA, Dahl DC, Silkensen JR, Sahadevan M, Snyder JJ. Hypertension after kidney transplantation. Am J Kidney Dis. 2004 Jun;43(6):1071-81. doi: 10.1053/j.ajkd.2004.03.013. PMID 15168388
- [Background] Paoletti E, Gherzi M, Amidone M, Massarino F, Cannella G. Association of arterial hypertension with renal target organ damage in kidney transplant recipients: the predictive role of ambulatory blood pressure monitoring. Transplantation. 2009 Jun 27;87(12):1864-9. doi: 10.1097/TP.0b013e3181a76775. PMID 19543066
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597